CLINICAL TRIAL: NCT03764059
Title: A Randomized Multicenter Two-Arm Clinical Study to Evaluate the Safety and Efficacy of Filtek™ Bulk Fill Posterior Restorative in Class I and II Restorations
Brief Title: Clinical Study of Filtek™ Bulk Fill Posterior Restorative in Class I and II Restorations
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: 3M (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MDI0102
Record Dates: First submitted 2018-12-03; First posted 2018-12-04 (Actual); Results first posted 2023-07-21 (Actual); Last update posted 2023-07-21 (Actual); Status verified 2023-07

CONDITIONS: Dental Caries Class I; Dental Caries Class II
Keywords: dental restorative; Composite posterior restorative

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Investigational device/experimental group: Filtek™ Bulk Fill Posterior Restorative (Experimental): The investigational device, Filtek™ Bulk Fill Posterior Restorative, was used for class 1 or 2 restorative in experimental group. The clinical assessments were performed immediately after restoration and included restoration retention/fracture, marginal fracture, anatomic form/marginal integrity, proximal contact, color match, surface texture/roughness, staining, marginal discoloration/secondary caries and pulp vitality.
  Subjects returned to the site for follow up visits at 1 week and 1 year postoperative for the same clinical assessments.
  Interventions: Device: Filtek™ Bulk Fill Posterior Restorative
- Control device/control group: Filtek™ Z350XT Universal Restorative (Active Comparator): The control device, Filtek™ Z350XT Universal Restorative, which was approved by CFDA in 2010 and has been in the market for 5 years with some validated clinical data, was used for class 1 or 2 restorative in control group. The clinical assessments were performed immediately after restoration and included restoration retention/fracture, marginal fracture, anatomic form/marginal integrity, proximal contact, color match, surface texture/roughness, staining, marginal discoloration/secondary caries and pulp vitality.
  Subjects returned to the site for follow up visits at 1 week and 1 year postoperative for the same clinical assessments.
  Interventions: Device: Filtek™ Z350XT Universal Restorative

INTERVENTIONS:
Device: Filtek™ Bulk Fill Posterior Restorative — The subjects were assigned to either the investigational device (Filtek™ Bulk Fill Posterior Restorative) or the control device (Filtek™ Z350XT Universal Restorative) per web-based randomization system.
  Arms: Investigational device/experimental group: Filtek™ Bulk Fill Posterior Restorative
Device: Filtek™ Z350XT Universal Restorative — The subjects were assigned to either the investigational device (Filtek™ Bulk Fill Posterior Restorative) or the control device (Filtek™ Z350XT Universal Restorative) per web-based randomization system.
  Other Names: Filtek™ Supreme Ultra Universal Restorative; Filtek™ Supreme XTE Universal Restorative; Filtek™ Ultimate Universal Restorative
  Arms: Control device/control group: Filtek™ Z350XT Universal Restorative

SUMMARY:
Purpose of the Study:This study was to evaluate the 1 week, 1 year safety and effectiveness of dental composite resin (Filtek™ Bulk Fill Posterior Restorative) in restoring Class I and II dental cavities in posterior teeth.

DETAILED DESCRIPTION:
This was a randomized, two- arm, non-inferiority study to evaluate the safety and clinical performance of resin composite, Filtek™ Bulk Fill.

Test apparatus: Apparatus for Test: Filtek™ Bulk Fill Posterior Restorative Apparatus for Control: 3M™ ESPE™ Filtek™ Z350XT, was approved by CFDA in 2010 and had been in the market for 5 years with some validated clinical data.

Sample Size of Subjects: Two-hundred forty (240) patients were expected to be recruited into the study and were randomly assigned to the test group and the control group according to the ratio of 1: 1; thus the number of cases in each group was 120. Finally, a total of 240 subjects were randomly enrolled in the study, including 120 subjects in the test group and 120 subjects in the control group, which met the required sample size.

The study consisted of screening period (initial screening visit, post-preparation screening visit), 1-week follow-up visit and 1-year follow-up visit, during which all the tests required in the protocol would be conducted to select the subjects meeting the criteria for inclusion. The examination and evaluation of the initial screening period were supposed to be completed within 0.5 days. Then investigators would make an appointment with the subjects eligible for the initial screening for cavity preparation and tooth filling, the required time of which depended on the complexity of the tooth problem and would be completed within 0.5 days. Immediate evaluation of relevant indicators were offered to the subjects who were selected and qualified after preparation and patients with qualified score would continue to have the 1-week and 1-year follow-up visits.

Subjects were randomly assigned to either the test group (Filtek™ Bulk Fill Posterior Repository) or the control group (Filtek™ Z350XT) in a central random manner, using the corresponding test product or control product to fill and restore posterior teeth defects (class I or class II cavities).

Since all investigators were required to operate according to instructions, it was clear to them which product a subject was given. However, subjects and clinical evaluators were blinded regarding whether the test product (Filtek™ Bulk Fill Posterior Repository) or the control product (Filtek™ Z350XT) was used by the subjects.

Immediately after restoration placement, at 1 week and 1 year postoperative, two or three clinical evaluators from each site performed the clinical assessment (the third more senior evaluator performed the assessment and determination if the first two evaluators were not in agreement) per China Technical Instruction and Guidance of Resin Composite Restoration Material For CFDA Registration (Technical Instruction and Guidance in short). The clinical acceptable rate of the restoration at 1 year was the primary endpoint in this study.

AE/SAE were collected to evaluate the safety of Filtek™ Bulk Fill. Based on the assessment result, if the clinical acceptance rate of the two groups achieved the clinical acceptable rate defined in the protocol, it indicated that Filtek™ Bulk Fill was efficacious for class 1 and II restorations.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female,18 to 70 years old (including 18 and 70 years)
2. Good health, no significant systemic disease;
3. Normal opening degree;
4. Molar (preferred) or premolar teeth
5. Cavity type with belongs to any of the following： 1) Class I, including the failed class I restoration which require to be repaired.; 2) Class II, including premolar and molar except the second molar (the failed class II restoration which require to be repaired is also included), and the gingival wall of cavity is above the free gingival margin coronally; 3) Class II cavity on the second molar when the third molar exists, and the gingival wall of cavity is above the free gingival margin coronally; 4) Class II, MO or MOD cavity on the second molar when the third molar does not exist (the failed class II restoration which require to be repaired is also included), and the gingival wall of cavity is above the free gingival margin coronally;
6. Cavity size: the buccolingual diameter of cavity is no less than the 1/3 and of the buccolingual cusp distance;
7. Occlusion with natural teeth;
8. Cavity depth: no less than 1/2 of dentin with a normal pulp status;
9. Be able to understand informed consent and to provide written inform consent ;
10. Be in good compliance with the protocol and willing to return to the site for follow up visits .

Exclusion Criteria:

1. Allergy to multiple medicines; allergy to resin or other polymer material;
2. Acute caries, severe periodontitis, salivary glands malfunction, dysfunction/disorder of TMJ (temporomandibular joint);
3. Poor oral hygiene, DMTF:18-34y >4, 35-70y >5;
4. Teeth with abnormal staining ;
5. Pathological abrasion (e.g. bruxism, clenching), acid corrosion, cracked-teeth and other non-caries diseases.
6. Abnormal occlusion;
7. Severe systemic or mental disorders;
8. Pregnant or intended to be pregnant (pregnant test is positive ) or breast feeding women;
9. Cavity do not meet the criteria based on the investigator's judgement;
10. Resin Composite is not an appropriate restoration for the subject
11. Pulp exposure or bottom of cavity is nearly close to the pulp;
12. Subjects who is not able to return for the one year follow-up visit because of going abroad or other reasons;
13. Subject is enrolled in other studies on investigational drug or device
14. Cannot tolerate rubber dam isolation. -

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2017-10-17 (Actual); Primary Completion 2019-11-14 (Actual); Study Completion 2019-11-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoyan Wang, Director, Principal Investigator — Endodontics department of Peking University hospital of stomatology
Locations (3):
- China (3):
  - Beijing Stomatology Hospital of Capital Medical University, Beijing, Beijing Municipality
  - Peking University Hospital of Stomatology, Beijing, Beijing Municipality
  - Hospital of Stomatology Wuhan University, Wuhan, Hubei

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Investigational Device/Experimental Group: Filtek™ Bulk Fill Posterior Restorative | Control Device/Control Group: Filtek™ Z350XT Universal Restorative
Started | 120 | 120
Completed | 120 | 120
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Interventional: The experimental group (Filtek Bulk fill posterior restoration) .After restoration,subjects will return to site for follow up visit at 1 week and 1 year postoperative for further clinical assessments.
  Filtek bulk fill posterior restoration: The subjects will be assigned to either the investigational product (Filtek Bulk ) or the control product (Z350XT) per web-based randomization system.
  Immediately after restoration placement, at 1 week and 1 year postoperative, two evaluators from each site will perform an independent clinical assessment.
- Observational: The control group (Filtek™ Z350XT Universal Restorative which was approved by CFDA in 2010 and has been in the market for 5 years with some validated clinical data).After restoration,subjects will return to the site for follow up visits at 1 week and 1 year postoperative for for further clinical assessments.
  Filtek™ Z350XT Universal Restorative: Filtek™ Z350XT Universal Restorative (Z350 XT) will serve as the control in this study.
- Total: Total of all reporting groups
Arm/Group | Interventional | Observational | Total
Number analyzed (Participants) | 120 | 120 | 240
Age, Continuous [Mean (Standard Deviation); unit: years] | 27.97 (6.65) | 28.12 (7.76) | 28.05 (10.22)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 84 | 81 | 165
  Male | 36 | 39 | 75
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Clinical diagnosis of caries [Number; unit: participants] | 119 | 120 | 239

OUTCOME MEASURES:

1. Primary Outcome: Clinical Acceptance Rate of Restoration at 1 Year After Replacement
Description: According to Clinical Trial Guideline for Polymer-based Dental Restorative Materials (YY/T 0990-2015), the clinically acceptable definition of restoration at 1 year after replacement was as follows: The retention and fracture score of restoration at 1 year after replacement was A; the marginal fracture, the appearance and the marginal adaptationof restoration was A or B.
Time Frame: 1 Year after restoration
Measure: Count of Participants; unit: Participants
Arm/Group | Investigational Device/Experimental Group: Filtek™ Bulk Fill Posterior Restorative | Control Device/Control Group: Filtek™ Z350XT Universal Restorative
Number analyzed (Participants) | 120 | 120
Participants
  Acceptable restoration | 120 | 119
  unacceptable restoration | 0 | 1
Statistical Analysis 1: Comparison: Investigational Device/Experimental Group: Filtek™ Bulk Fill Posterior Restorative vs Control Device/Control Group: Filtek™ Z350XT Universal Restorative; Test type: Non-Inferiority — The test for non-inferiority is based on a 95% CI of the difference between the investigational and control groups with respect to the rate of clinically acceptable restorations at 1-year post placement. The non-inferiority margin was 7%. To establish non-inferiority the lower limit has to be > -7%; p < 0.0001, Cochran-Mantel-Haenszel; Risk Difference (RD) = 4.2, 95% CI 2-sided [- 0.6 to 9.2]

ADVERSE EVENTS:
Time Frame: Adverse Events (AEs) and Serious Adverse Events (SAEs) were collected from enrollment through study completion, an average of 1 year per participant.
Arm/Group | Investigational Device/Experimental Group: Filtek™ Bulk Fill Posterior Restorative | Control Device/Control Group: Filtek™ Z350XT Universal Restorative
All-Cause Mortality (participants affected / at risk) | 0/120 | 0/120
Serious Adverse Events (participants affected / at risk) | 0/120 | 0/120
Other Adverse Events (participants affected / at risk) | 45/120 | 36/120
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Investigational Device/Experimental Group: Filtek™ Bulk Fill Posterior Restorative (N=120) | Control Device/Control Group: Filtek™ Z350XT Universal Restorative (N=120)
Upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 5 | 8
Non-target caries (Gastrointestinal disorders) | 20 | 5
Post-operative tooth sensitivity (Gastrointestinal disorders) | 8 | 3
Impacted wisdom teeth (Gastrointestinal disorders) | 6 | 7
Wisdom tooth extraction (Gastrointestinal disorders) | 3 | 0
Acne (Skin and subcutaneous tissue disorders) | 0 | 2
Periodontitis (Gastrointestinal disorders) | 0 | 1
Irregular dentition (Gastrointestinal disorders) | 1 | 2
Tooth sensitivity during operation (Gastrointestinal disorders) | 0 | 1
Kidney stone (Renal and urinary disorders) | 0 | 1
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 | 1
Chronic periodontitis (Gastrointestinal disorders) | 1 | 2
Chronic periapical periodontitis (Gastrointestinal disorders) | 0 | 1
Plaque-induced gingivitis (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 1
Gum bleeding on the target side (Gastrointestinal disorders) | 1 | 0
Gum pain on the target side (Gastrointestinal disorders) | 1 | 0
Mild redness and swelling of gingival margin on the target side (Gastrointestinal disorders) | 1 | 1
Pain of buccal mucosa of target teeth (Gastrointestinal disorders) | 0 | 1
Mucosal ulceration of target teeth (Gastrointestinal disorders) | 1 | 0
Radiolucent area of root tip of target teeth (Gastrointestinal disorders) | 0 | 1
Malaise of occlusion of target teeth (Gastrointestinal disorders) | 1 | 1
Spontaneous discomfort of target teeth (Gastrointestinal disorders) | 1 | 0
Edge caries of non-target teeth (Gastrointestinal disorders) | 1 | 0
Non-target residual root (Gastrointestinal disorders) | 0 | 1
Falling of filling material of non-target teeth (Product Issues) | 1 | 0
Pericoronitis of non-target teeth (Gastrointestinal disorders) | 3 | 1
Secondary Caries of non-target teeth (Gastrointestinal disorders) | 1 | 0
Secondary Caries of non-target teeth (after endodontic treatment) (Gastrointestinal disorders) | 1 | 1
Reversible pulpitis of non-target teeth (Gastrointestinal disorders) | 1 | 0
Chronic pulpitis of non-target teeth (Gastrointestinal disorders) | 1 | 0
Acute attack of chronic pulpitis of non-target teeth (Infections and infestations) | 0 | 1
Non-target caries, gingivitis (Gastrointestinal disorders) | 1 | 0
Sensitivity of non-target teeth after operation (Gastrointestinal disorders) | 0 | 2
Microdontia of non-target teeth (Gastrointestinal disorders) | 1 | 0
Wedge-shaped defect of non-target teeth (Gastrointestinal disorders) | 0 | 2
Pulpitis of non-target teeth (Gastrointestinal disorders) | 1 | 0
Dental defect of non-target teeth (Gastrointestinal disorders) | 1 | 1
Gingival ulcer of non-target teeth (Gastrointestinal disorders) | 1 | 0
Treatment of non-target teeth (Surgical and medical procedures) | 1 | 0
Mild redness and swelling of gingival margin of non-target teeth (Gastrointestinal disorders) | 2 | 0
Recurrent oral ulcer (Gastrointestinal disorders) | 0 | 1
Generalized chronic periodontitis (Gastrointestinal disorders) | 1 | 0
Acute laryngitis (Infections and infestations) | 1 | 0
Pain in the injection point of buccal anesthetics (Gastrointestinal disorders) | 1 | 0
Redness and swelling of gingiva near middle palatal side (Gastrointestinal disorders) | 1 | 0
Coughing (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Chestnut eruption (Skin and subcutaneous tissue disorders) | 1 | 0
Other Treatments (Surgical and medical procedures) | 0 | 1
Gingival margin of palatine side injured by rubber dam (Injury, poisoning and procedural complications) | 1 | 0
Gingival edema (Gastrointestinal disorders) | 1 | 0
Right ankle fracture (Musculoskeletal and connective tissue disorders) | 1 | 0
Hordeolum (Eye disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2018-08-20): https://cdn.clinicaltrials.gov/large-docs/59/NCT03764059/Prot_000.pdf
  • Statistical Analysis Plan (2020-03-03): https://cdn.clinicaltrials.gov/large-docs/59/NCT03764059/SAP_001.pdf